CLINICAL TRIAL: NCT05118139
Title: CSD201203: A Study to Determine Subject Puffing Patterns of a Non-cylindrical, Closed, Electronic Nicotine Delivery System at Three Nicotine Concentrations in an Ambulatory Setting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RAI Services Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CSD201203
Record Dates: First submitted 2021-11-01; First posted 2021-11-11 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Smoking; Tobacco Use; Electronic Cigarette Use
MeSH Terms: conditions — Smoking; Tobacco Use; Vaping

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 1.5% nicotine cartridges (Experimental): Subjects will self-assign to one of 7 flavor variants of 1.5% ENDS products based on their preferred flavor.
  Interventions: Other: P1211216; Other: P1213416; Other: P1213716; Other: P1213616; Other: P1213816; Other: P1211916; Other: P1210016
- 2.4% nicotine cartridges (Experimental): Subjects will self-assign to one of 2 flavor variants of 2.4% ENDS products based on their preferred flavor.
  Interventions: Other: P1211217; Other: P1213417
- 5% nicotine cartridges (Experimental): Subjects will self-assign to one of 7 flavor variants of 5% ENDS products based on their preferred flavor.
  Interventions: Other: P1211222; Other: P1213422; Other: P1213722; Other: P1213622; Other: P1213822; Other: P1211922; Other: P1210022

INTERVENTIONS:
Other: P1211216 — Flavor variant P1211216 of a 1.5% nicotine ENDS product
  Arms: 1.5% nicotine cartridges
Other: P1213416 — Flavor variant P1213416 of a 1.5% nicotine ENDS product
  Arms: 1.5% nicotine cartridges
Other: P1213716 — Flavor variant P1213716 of a 1.5% nicotine ENDS product
  Arms: 1.5% nicotine cartridges
Other: P1213616 — Flavor variant P1213616 of a 1.5% nicotine ENDS product
  Arms: 1.5% nicotine cartridges
Other: P1213816 — Flavor variant P1213816 of a 1.5% nicotine ENDS product
  Arms: 1.5% nicotine cartridges
Other: P1211916 — Flavor variant P1211916 of a 1.5% nicotine ENDS product
  Arms: 1.5% nicotine cartridges
Other: P1210016 — Flavor variant P1210016 of a 1.5% nicotine ENDS product
  Arms: 1.5% nicotine cartridges
Other: P1211217 — Flavor variant P1211217 of a 2.4% nicotine ENDS product
  Arms: 2.4% nicotine cartridges
Other: P1213417 — Flavor variant P1213417 of a 2.4% nicotine ENDS product
  Arms: 2.4% nicotine cartridges
Other: P1211222 — Flavor variant P1211222 of a 5% nicotine ENDS product
  Arms: 5% nicotine cartridges
Other: P1213422 — Flavor variant P1213422 of a 5% nicotine ENDS product
  Arms: 5% nicotine cartridges
Other: P1213722 — Flavor variant P1213722 of a 5% nicotine ENDS product
  Arms: 5% nicotine cartridges
Other: P1213622 — Flavor variant P1213622 of a 5% nicotine ENDS product
  Arms: 5% nicotine cartridges
Other: P1213822 — Flavor variant P1213822 of a 5% nicotine ENDS product
  Arms: 5% nicotine cartridges
Other: P1211922 — Flavor variant P1211922 of a 5% nicotine ENDS product
  Arms: 5% nicotine cartridges
Other: P1210022 — Flavor variant P1210022 of a 5% nicotine ENDS product
  Arms: 5% nicotine cartridges

SUMMARY:
This is a multi-center, open-label, parallel, three-study-group investigation to evaluate the puffing patterns of healthy adult consumers of tobacco products switching from a usual brand (UB) Electronic Nicotine Delivery Systems (ENDS) product to the ENDS Investigational Product (IP), over a 9-day ambulatory period.

DETAILED DESCRIPTION:
Potential subjects may complete a pre-screening interview and will complete a Screening Visit to assess their eligibility. Based on meeting eligibility requirements, subjects will be enrolled into the study either on the same day of their Screening Visit or return to the clinic on another day to complete the Enrollment Visit.

Subjects will be assigned to one of three nicotine concentrations of the IP based on their scheduled Enrollment Visit to the clinic. Once enrolled, the subjects will be assigned to one of the flavor variants of the IP after sampling or trying flavors, within the assigned nicotine concentration, and determining which flavor that they would like to use for the length of the study. Once a particular flavor group has reached full enrollment, that flavor will no longer be available for sampling and selection. Subjects will be instructed not to use their UB ENDS products during the study.

At the Enrollment Visit, subjects will be provided a Power Unit, Cartridges for their assigned product, a Product Use and Behavior (PUB) instrument, and an electronic device. The electronic device will have the PUB application installed for topography data capture and PUB data transmission. Based upon their UB ENDS usage, subjects will be given a sufficient amount of their assigned IP cartridges.

Subjects will be instructed to use their assigned IP in place of their UB ENDS during the 9-day study period (including a 2-day IP acclimation period followed by a 7-day product use evaluation period). Subjects will be allowed to use non-ENDS tobacco- or nicotine-containing products according to their normal use pattern. The PUB instrument will collect puffing topography data throughout the product use period.

At the end of the 2-day IP acclimation period, subjects will receive a phone call from the clinic to assess IP compliance and to ensure that they are not using their UB ENDS. During the following Days 3-9 evaluation period, subjects will receive a phone call to remind them of guidelines for using their assigned IP and to document adverse events (AEs).

At the conclusion of the 9-day ambulatory period, the subjects will return to the clinic, return the Power Unit, any associated Accessory USB Charger, all used and unused IP cartridges, the corresponding PUB instrument and its charger, and the electronic device. Each subject will complete all End of Study procedures including completing the Product Evaluation Scale (PES) questionnaire and two additional questionnaires to assess the degree of overall product liking and intention to use the product. The subjects will then be discharged from the study.

ELIGIBILITY:
Inclusion Criteria:

1. Able to read, understand, and willing to sign an informed consent form (ICF) and complete questionnaires written in English.
2. Generally healthy male or female adults, ≥ 21 years of age, inclusive, at the time of consent.
3. Positive urine cotinine test at the Screening Visit.
4. Non-cylindrical, cartridge-based, closed-system ENDS are the primary form of tobacco- or nicotine-containing products used within 30 days of the Screening Visit. Subjects may be users of other tobacco- or nicotine-containing products. If the subject is a dual/poly user of tobacco- or /nicotine-containing products then the subject must self-report that a non-cylindrical, cartridge-based, closed-system ENDS is their primary product.
5. Must have used 2 or more cartridges per week over the last 30 days. Brief periods of abstinence due to illness, quit attempt (prior to 30 days of the Screening Visit), or clinical study participation (prior to 30 days of the Screening Visit) will be allowed at the discretion of the Principal Investigator (PI).
6. Females must be willing to use a form of contraception acceptable to the PI from the time of signing the ICF until the end of the study.
7. Must be willing to use the assigned IP and only the assigned flavor as their exclusive source of ENDS use for the full duration of the 9-day ambulatory period. Use of other non-ENDS tobacco- or nicotine-containing products will be permitted during the ambulatory period.
8. Must have familiarity with modern electronic devices such as an IOS/Android smart phone or tablet computer ("tablet") and be willing to be provided with an electronic device, that allows for both Bluetooth connectivity and internet connectivity. Must be willing to use an application on the electronic device and keep the application active for the length of the study
9. Able to safely perform the required study procedures, as determined by the PI.

Exclusion Criteria:

1. Presence of clinically significant uncontrolled cardiovascular, pulmonary, renal, hepatic, endocrine, gastrointestinal, psychiatric, hematological, neurological disease, or any other concurrent disease or medical condition that, in the opinion of the PI, makes the study subject unsuitable to participate in this clinical study.
2. History of or presence of diabetes.
3. Systolic blood pressure of > 160 mmHg or a diastolic blood pressure of > 95 mmHg, measured after being seated for five minutes, with exceptions at the PI's discretion.
4. Scheduled treatment for asthma currently or within the past consecutive 12 months prior to the Screening Visit. As-needed treatment, such as inhalers, may be included at the PI's discretion pending approval from the Medical Monitor.
5. Any history of cancer, except for primary cancers of skin such as localized basal cell/squamous cell carcinoma that has been surgically and/or cryogenically removed.
6. Use of any medication or substance that aids in smoking cessation, including but not limited to any nicotine replacement therapy (NRT, e.g., nicotine gum, lozenge, patch), varenicline (Chantix®), bupropion (Wellbutrin®, Zyban®), or lobelia extract within (≤) 30 days prior to the signing the ICF.
7. Participation in another clinical trial within (≤) 30 days prior to signing the ICF unless allowed at the discretion of the Principal Investigator (PI). The 30-day window for each subject will be derived from the date of the last study event in the previous study to the time of signing the ICF in the current study.
8. Females who have a positive pregnancy test, or who are pregnant, are breastfeeding, or intend to become pregnant during the course of the study.
9. Individuals ≥ 35 years of age currently using systemic, estrogen-containing contraception or hormone replacement therapy.
10. A positive urine drug screen without evidence of prescribed corresponding concomitant medication(s) at the Screening or Enrollment Visits.
11. Postpones a decision to quit using tobacco- or nicotine-containing products in order to participate in this study or a previous attempt within (≤) 30 days prior to signing the ICF.
12. Drinks more than 21 servings of alcoholic beverages per week or has a positive test for alcohol result at the Screening or Enrollment Visits.
13. Employed by a tobacco- or nicotine-manufacturing company, the study site, or handles tobacco- or nicotine-containing products as part of their job.
14. Determined by the PI to be inappropriate for this study.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2022-02-11 (Actual); Primary Completion 2022-07-30 (Actual); Study Completion 2022-07-30 (Actual)

PRIMARY OUTCOMES:
Puff duration | Final 7 days of data collection
  Average puff duration
Number of puff per day | Final 7 days of data collection
  Average number of puffs per day

CONTACTS AND LOCATIONS:
Overall Officials: Gary Dull, PhD, Study Director — RAIS
Locations (4):
- United States (4):
  - Clinical Research Atlanta, Stockbridge, Georgia
  - AMR Lexington, Lexington, Kentucky
  - Accellacare Hickory, Hickory, North Carolina
  - High Point Clinical Trials Center, High Point, North Carolina

IPD SHARING:
Plan to Share IPD: No